CLINICAL TRIAL: NCT03771807
Title: A Single-center, Placebo Controlled Study to Investigate the Efficacy of a Nutritional Supplement on Skin Health in Generally Healthy Adults
Brief Title: Efficacy of a Nutritional Supplement on Skin Health in Generally Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Dermatology Consulting Services, High Point NC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 18-PHX-0002
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Skin Health

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo & facial cleansing (Placebo Comparator): Maltodextrin and food coloring
  Subjects will clean the right side of their face with a cosmetic instrument daily
  Interventions: Other: Placebo; Other: Facial cleansing
- Beauty From Within & facial cleansing (Active Comparator): Study Product contains collagen hydrolysate, ceramide wheat extract oil and lutein
  Subjects will clean the right side of their face with a cosmetic instrument daily
  Interventions: Dietary Supplement: Beauty From Within; Other: Facial cleansing

INTERVENTIONS:
Dietary Supplement: Beauty From Within — one scoop of product mixed in 8-16 ounces of water consumed once daily
  Arms: Beauty From Within & facial cleansing
Other: Placebo — one scoop of product mixed in 8-16 ounces of water consumed once daily
  Arms: Placebo & facial cleansing
Other: Facial cleansing — All subjects will use a cosmetic instrument to clean on one half of their face daily

SUMMARY:
Consumption of dietary supplements has been found to modulate skin health. Individual ingredients such as collagen peptides, lutein and ceramides have been shown to improve skin health. Collagen peptides have been shown to clinically improve skin texture, decrease area of skin ultraviolet damage, increase skin hydration, and improve visible skin results such as hydration, elasticity, wrinkles and roughness. Lutein has been demonstrated to increase skin radiance, protect skin from ultraviolet light, and increase skin hydration. Ceramides derived from wheat have been shown to improve skin texture, increase skin hydration and improve visible skin attributes such as hydration, elasticity, and wrinkles. This study will have subjects consuming a nutritional supplement or placebo daily for 90 days to see if there is an effect on skin health. This study will also have the subjects using a facial cleansing device, which has been shown to improve skin health, on half of their face to determine if there is a synergistic effect between dietary supplement and cleansing device. It is believed, this mixture of collagen peptides, lutein and ceramides has not been studied and the study sponsor hypothesize that this blend of ingredients will have a positive impact on skin health.

DETAILED DESCRIPTION:
Visit 1 Screening (day -30 to -1): Subjects will be given a copy of the informed consent document. They will be given ample time to read and formulate questions prior to reviewing the document with study staff. The consent form will be reviewed with the subject and questions will be answered. The subject will provide written consent prior to starting any study related assessments. The study staff will collect the following information during this visit:

* Review medical history
* Review concomitant medications
* Measure height, weight, BMI, heart rate, blood pressure
* Review inclusion/exclusion criteria

If the subject meets inclusion/exclusion criteria they will complete the following study assessments.

* Skin examination
* Investigator facial clinical grading
* Corneometry of both sides of the face and one forearm
* Colorimeter of both sides of the face and one forearm
* Elasticity of both sides of the face
* Carotenoid scan of left hand
* AGE reader of left forearm
* Digital photo of face

Visit 2 Baseline (day 0): Subjects will return to the research site for baseline visit approximately 30 days after their screening visit. Subjects will undergo assessments to determine that they continue to meet inclusion/exclusion criteria. Subjects who are eligible will be enrolled into the study and assigned a randomization number and study product. The following assessments will be completed during this visit:

* Measure weight, BMI, heart rate, blood pressure
* Investigator facial clinical grading
* Subject facial grading
* Corneometry of both sides of the face and one forearm
* Colorimeter of both sides of the face and one forearm
* Elasticity of both sides of the face
* Carotenoid scan of left hand
* AGE reader of left forearm
* 10ml Blood draw (Chemistry and CBC)
* Digital photo of face
* UV Radiation of buttocks (1MED, 2MED, 3MED)

Visit 3 Baseline + 24hrs (day 1): Subjects will return to the research site approximately 24hrs after their baseline visit. The following assessments will be completed during this visit:

* Digital photograph of irradiated buttock site
* Dermospectrophotometer of irradiated site
* Dispense 2 months of assigned study product
* Dispense skin cleansing machine and provide instruction on daily use to the right half of their face only

Visit 4 (day 30 +5 days): Subjects will return at approximately 30 days after their baseline visit. Unused study product will be collected and compliance will be calculated. The following assessments will be completed:

* Investigator facial clinical grading
* Subject facial grading
* Corneometry of both sides of the face and one forearm
* Colorimeter of both sides of the face and one forearm
* Elasticity of both sides of the face
* Carotenoid scan of left hand
* AGE reader of left forearm
* Adverse events will be collected by asking if the subject has experienced any changes in their health
* Return unused study product and dispense enough assigned study product to make it through next study visit

Visit 5 (day 60 +5 days): Subjects will return at approximately 60 days after their baseline visit. Unused study product will be collected and compliance will be calculated. The following assessments will be completed:

* Investigator facial clinical grading
* Subject facial grading
* Corneometry of both sides of the face and one forearm
* Colorimeter of both sides of the face and one forearm
* Elasticity of both sides of the face
* Carotenoid scan of left hand
* AGE reader of left forearm
* Adverse events will be collected by asking if the subject has experienced any changes in their health
* Return unused study product and dispense enough assigned study product to make it through next study visit

Visit 6 (day 90 +5 days): Subjects will return at approximately 90 days after their baseline visit. Unused study product will be collected and compliance will be calculated. The following assessments will be completed:

* Measure weight, BMI, heart rate, blood pressure
* Investigator facial clinical grading
* Subject facial grading
* Corneometry of both sides of the face and one forearm
* Colorimeter of both sides of the face and one forearm
* Elasticity of both sides of the face
* Carotenoid scan of left hand
* AGE reader of left forearm
* 10ml Blood draw (Chemistry and CBC)
* Digital photo of face
* UV Radiation of buttocks (1MED, 2MED, 3MED)
* Collect skin cleansing machine
* Adverse events will be collected by asking if the subject has experienced any changes in their health

Visit 7 (24 hours after visit 6): Subjects will return to the research site approximately 24hrs after visit 6. The following assessments will be completed during this visit:

* Digital photograph of irradiated buttock site
* Dermospectrophotometer of irradiated site

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 40 - 60 years of age
2. Individuals must present with stable moderate signs of aging that does not change between the screening visit and the baseline visit 4 weeks later
3. Subject is willing and able to participate in all aspects of the study
4. Individuals must sign informed consent, photo release consent and confidentiality agreement
5. Subject has a BMI > 19 and < 32
6. Subject must be on a stable dose of chronic use medications for at least 3 months prior to study participation
7. Subject who, in the opinion of the investigator, are free of any medical condition(s) that may interfere with study participation or affect study measures

Exclusion Criteria:

1. Individuals that are being treated for cancer or have a history of facial skin cancer
2. Individuals with sunburn, moderate to pronounced suntan, uneven skin tones, tattoos, scares or other disfiguration, dilated vessels or other conditions on the test area that might influence the test results
3. Any disease or condition of the skin that the investigator deems inappropriate for participation, including rosacea, eczema, psoriasis, and atopic dermatitis
4. Individuals currently taking medications which in the opinion of the investigator may interfere with the study. This would include but not be limited to all oral corticosteroids, use of anti-inflammatory drugs more than 14 consecutive days, immunosuppressive drugs or antihistamine medications (steroid nose drops and/or eye drops are permitted), hormone replacement therapy and insulin, antibiotics or other topical drugs at the test sites
5. Individuals with uncontrolled metabolic diseases such as diabetes (type I and II), hypertension, hyperthyroidism or hypothyroidism, severe chronic asthma, immunological disorders such as HIV, AIDS and systemic lupus erythematosus or mastectomy for cancer involving removal of lymph nodes
6. Subject is taking skin, nail, and hair health promoting supplement orally (including products containing collagen and carotenoids)
7. Women known to be pregnant, nursing, or planning to become pregnant
8. Individuals participating in other facial clinical trials
9. Individuals who have routinely used alpha-hydroxy-acid (AHA) or a beta-hydroxy-acid (BHA) containing product within two weeks of baseline visit or Retin-A®, Retin-A Micro®, Renova®, Differin®, Avita®, Tazorac®, or Soriatane® within one month of baseline visit or have taken Accutane® within one year of baseline visit. Individuals who have used Retinol in the last six months prior to baseline visit
10. Individuals with inflammatory acne lesions (i.e., papules, pustules, cysts, nodules) at the test site
11. Individuals who have had chemical peels or dermabrasion within the last six months prior to baseline visit
12. Individuals who have sun tanned (sun or tanning beds) in the nude within the past 1 year prior to baseline visit
13. Excessive alcohol use (>2 drinks per day)
14. Subject is a current smoker or quit less than 3 years from screening visit
15. History of substance abuse

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Skin Health (lines) | baseline, day 30, day 60, and day 90
  Change from baseline in investigator and subject facial grading of lines (using a scale 0=none, 1=minimal, 2=mild, 3=moderate, 4=severe) at days 30, 60, and 90 using Mann Whitney two tailed assessment for nonparametric data
Skin Health (firmness) | baseline, day 30, day 60, and day 90
  Change from baseline in investigator and subject facial grading of firmness (using a scale 0=none, 1=minimal, 2=mild, 3=moderate, 4=severe) at days 30, 60, and 90 using Mann Whitney two tailed assessment for nonparametric data
Skin Health (radiance) | baseline, day 30, day 60, and day 90
  Change from baseline in investigator and subject facial grading of radiance (using a scale 0=none, 1=minimal, 2=mild, 3=moderate, 4=severe) at days 30, 60, and 90 using Mann Whitney two tailed assessment for nonparametric data
Skin Health (texture) | baseline, day 30, day 60, and day 90
  Change from baseline in investigator and subject facial grading of texture (using a scale 0=none, 1=minimal, 2=mild, 3=moderate, 4=severe) at days 30, 60, and 90 using Mann Whitney two tailed assessment for nonparametric data
Skin Health (overall) | baseline, day 30, day 60, and day 90
  Change from baseline in investigator and subject facial grading overall (using a scale 0=none, 1=minimal, 2=mild, 3=moderate, 4=severe) at days 30, 60, and 90 using Mann Whitney two tailed assessment for nonparametric data

SECONDARY OUTCOMES:
Cellular protection of the skin as determined by dermospectrophotometer of UV irradiated site | baseline, and day 91
  Change from baseline in dermospectrophotometer at day 91 using Student T-test
Skin elasticity of face determined by cutometer | baseline, day 30, day 60, and day 90
  Change from baseline in skin elasticity at days 30, 60, and 90 using Student T-test
Ramen skin carotenoids score determined by carotenoid scan of left hand | baseline, day 30, day 60, and day 90
  Change from baseline in skin carotenoids at days 30, 60, and 90 using Student T-test
Benefits of facial cleansing in concurrence with dietary supplement | baseline, day 30, day 60, and day 90
  Determine if facial cleansing improves outcomes over dietary supplement use alone as determined by investigator assessment using a scale 0=none, 1=minimal, 2=mild, 3=moderate, 4=severe in lines, firmness, radiance, texture, and overall of both sides of the subjects face

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Dermatology Consulting Services, High Point NC
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bizot, V., E. Cestone, A. Michelotti and V. Nobile. Improving skin hydration and age-related symptoms by oral administration of wheat glucosylceramides and digalactosyl diglycerides: a human clinical study. Cosmetics 4(37): 2017
- [Background] Juturu V, Bowman JP, Deshpande J. Overall skin tone and skin-lightening-improving effects with oral supplementation of lutein and zeaxanthin isomers: a double-blind, placebo-controlled clinical trial. Clin Cosmet Investig Dermatol. 2016 Oct 7;9:325-332. doi: 10.2147/CCID.S115519. eCollection 2016. PMID 27785083
- [Background] Morganti P, Fabrizi G, Bruno C. Protective effects of oral antioxidants on skin and eye function. Skinmed. 2004 Nov-Dec;3(6):310-6. doi: 10.1111/j.1540-9740.2004.02420.x. PMID 15538079
- [Background] Palombo P, Fabrizi G, Ruocco V, Ruocco E, Fluhr J, Roberts R, Morganti P. Beneficial long-term effects of combined oral/topical antioxidant treatment with the carotenoids lutein and zeaxanthin on human skin: a double-blind, placebo-controlled study. Skin Pharmacol Physiol. 2007;20(4):199-210. doi: 10.1159/000101807. Epub 2007 Apr 19. PMID 17446716
- [Background] Proksch E, Schunck M, Zague V, Segger D, Degwert J, Oesser S. Oral intake of specific bioactive collagen peptides reduces skin wrinkles and increases dermal matrix synthesis. Skin Pharmacol Physiol. 2014;27(3):113-9. doi: 10.1159/000355523. Epub 2013 Dec 24. PMID 24401291
- [Background] Proksch E, Segger D, Degwert J, Schunck M, Zague V, Oesser S. Oral supplementation of specific collagen peptides has beneficial effects on human skin physiology: a double-blind, placebo-controlled study. Skin Pharmacol Physiol. 2014;27(1):47-55. doi: 10.1159/000351376. Epub 2013 Aug 14. PMID 23949208